CLINICAL TRIAL: NCT01105429
Title: Placebo-Controlled, Ascending Single-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BMS-820132 in Subjects With Type 2 Diabetes on Background Therapy of Metformin
Brief Title: Single Ascending Dose Study of BMS-820132 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MB122-002
Record Dates: First submitted 2010-04-13; First posted 2010-04-16 (Estimated); Last update posted 2011-03-09 (Estimated); Status verified 2010-11

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- BMS-820132 (0.3 mg) or Placebo (Active Comparator)
  Interventions: Drug: BMS-820132; Drug: Placebo
- BMS-820132 (1.0 mg) or Placebo (Active Comparator)
  Interventions: Drug: BMS-820132; Drug: Placebo
- BMS-820132 (3 mg) or Placebo (Active Comparator)
  Interventions: Drug: BMS-820132; Drug: Placebo
- BMS-820132 (10 mg) or Placebo (Active Comparator)
  Interventions: Drug: BMS-820132; Drug: Placebo
- BMS-820132 (30 mg) or Placebo (Active Comparator)
  Interventions: Drug: BMS-820132; Drug: Placebo
- BMS-820132 (75 mg) or Placebo (Active Comparator)
  Interventions: Drug: BMS-820132; Drug: Placebo
- BMS-820132 (150 mg) or Placebo (Active Comparator)
  Interventions: Drug: BMS-820132; Drug: Placebo
- BMS-820132 (300 mg) or Placebo (Active Comparator)
  Interventions: Drug: BMS-820132; Drug: Placebo
- BMS-820132 (TBD) or Placebo (Active Comparator)
  Interventions: Drug: BMS-820132; Drug: Placebo

INTERVENTIONS:
Drug: BMS-820132 — Oral Solution, Oral, 0.3 mg, once daily, 1 day
  Arms: BMS-820132 (0.3 mg) or Placebo
Drug: BMS-820132 — Oral Solution, Oral, 1.0 mg, once daily, 1 day
  Arms: BMS-820132 (1.0 mg) or Placebo
Drug: BMS-820132 — Oral Solution, Oral, 3 mg, once daily, 1 day
  Arms: BMS-820132 (3 mg) or Placebo
Drug: BMS-820132 — Oral Solution, Oral, 10 mg, once daily, 1 day
  Arms: BMS-820132 (10 mg) or Placebo
Drug: BMS-820132 — Oral Solution, Oral, 30 mg, once daily, 1 day
  Arms: BMS-820132 (30 mg) or Placebo
Drug: BMS-820132 — Oral Solution, Oral , 75 mg, once daily, 1 day
  Arms: BMS-820132 (75 mg) or Placebo
Drug: BMS-820132 — Oral Solution, Oral, 150 mg, once daily, 1 day
  Arms: BMS-820132 (150 mg) or Placebo
Drug: BMS-820132 — Oral Solution, Oral, 300 mg, once daily, 1 day
  Arms: BMS-820132 (300 mg) or Placebo
Drug: BMS-820132 — Capsule, Oral, (TBD), once daily, 2 days
  Arms: BMS-820132 (TBD) or Placebo
Drug: Placebo — Oral Solution, Oral, 0mg, once daily, 1 day
  Arms: BMS-820132 (0.3 mg) or Placebo; BMS-820132 (1.0 mg) or Placebo; BMS-820132 (10 mg) or Placebo; BMS-820132 (150 mg) or Placebo; BMS-820132 (3 mg) or Placebo; BMS-820132 (30 mg) or Placebo; BMS-820132 (300 mg) or Placebo; BMS-820132 (75 mg) or Placebo
Drug: Placebo — Capsule, Oral, (TBD), once daily, 2 days
  Arms: BMS-820132 (TBD) or Placebo

SUMMARY:
BMS-820132 is an investigational new drug being developed by BMS for treating Type 2 diabetes. The purpose of this study is to test the safety/tolerability (potential side effects) of single doses of the investigational new drug, as well as the amount of study drug in the blood, in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of childbearing potential (willing to use an acceptable method of contraception), or females of non-childbearing potential (i.e., post-menopausal or surgically sterile)
* Diagnosis of type 2 diabetes treated with metformin monotherapy on a stable regimen for at least 2 months
* Body Mass Index (BMI) of 18 to 40 kg/m2
* Fasting glucose in the range of 100-250 mg/dL
* Hemoglobin A1c (HbA1c) in the range of 6.5% -9.5%

Exclusion Criteria:

* Clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
* Any significant acute or chronic medical illness other than stable and well controlled hypertension, microalbuminuria, dyslipidemia, or depression
* Past history of diabetic ketoacidosis and/or C-peptide < 1.0 ng/mL, hyperosmolar nonketotic syndrome, lactic acidosis, or recurrent hypoglycemia
* Any major surgery within 4 weeks of study drug administration
* Any gastrointestinal surgery that could impact upon the absorption of study drug
* Smoking more than 10 cigarettes per day
* Recent drug or alcohol abuse
* Women who are pregnant or breastfeeding
* Positive urine screen for drugs of abuse
* Positive blood screen for hepatitis C antibody, hepatitis B surface antigen, or HIV-1, -2 antibody

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of the investigational drug, as assessed by adverse event monitoring, physical examinations, clinical laboratory determinations, electrocardiograms (ECG), and vital sign assessments | Within 5 days of study drug administration

SECONDARY OUTCOMES:
Exposure to the investigational drug and its metabolites | Within 2 days after study drug administration
Pharmacodynamic activity of the investigational drug on biomarkers | Within 2 days after study drug administration
Excretion of the investigational drug and metabolites from the body | Within 2 days after study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Profil Institute For Clinical Research, Inc. (Picr), Chula Vista, California
  - Clinical Pharmacology Of Miami Inc., Miami, Florida
  - Elite Research Institute, Miami, Florida

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx